CLINICAL TRIAL: NCT05925374
Title: Planning a Multi-Level Intervention to Reduce Substance Use Stigma in HIV Prevention and Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Loyola University Chicago (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin F. Madden, Assistant Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R34DA053758 (NIH); 5R34DA053758-03 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-29 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Social Stigma; Substance Use Disorders; HIV Infections; Physician-Patient Relations
Keywords: community-engaged research; Provider-based stigma; Structural stigma
MeSH Terms: conditions — Social Stigma; Substance-Related Disorders; HIV Infections

STUDY DESIGN:
Intervention Model Description: This study will pilot test a substance use training that aims to reduce professional stigma towards patients who use drugs. Participants will be professionals working in primary care settings, and all participants will receive the intervention (training). Their stigmatizing attitudes and intended/planned behaviors will be assessed immediately prior to the training and immediately after the training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training group (Experimental): Professionals working at a primary care site who has direct interaction with patients. They receive a one-time 2-hour interactive in-person training focused on improving care for patients who use drugs and reducing provider-based stigma. Their baseline attitudes and intended actions are compared to their post-intervention answers to questions in the same domains. Thus, the participants act as their own comparison group, where baseline answers are compared to post-intervention answers.
  Interventions: Behavioral: Substance use stigma training

INTERVENTIONS:
Behavioral: Substance use stigma training — The intervention is an interactive professional educational training that is designed to manipulate behavioral and normative beliefs in order to address bias and alter professional practices towards patients who use drugs.

SUMMARY:
This is a community-engaged research project that aims to identify and pilot test interventions that may reduce substance use stigma among professionals at primary care sites serving patients who might be exposed to HIV or are living with HIV. Our goal is to develop a multi-level substance use stigma intervention that leverages 1) education and 2) organizational policy to address structural drivers of stigma and the stigmatizing professional attitudes and behaviors that affect patients. Hypothesis: the results of the trial pilot research and are expected to provide scientific evidence demonstrating feasible and potentially effective substance use stigma reduction interventions that go beyond simple individual-level professional training. We plan to build on the data from this pilot trial study to then further test the multi-level intervention in another larger trial study with primary care organizations to determine whether the intervention addresses multiple complex drivers of substance use stigma that influence HIV prevention and care outcomes among people who use drugs.

DETAILED DESCRIPTION:
This planning project aims to develop and pilot test elements of a multi-level substance use stigma reduction intervention. This study builds on past research indicating educational interventions can meaningfully reduce provider stigma related to substance use by examining the extent to which educational interventions may be enhanced by organizational policies addressing structural drivers of stigma toward people who use drugs operating in the health sector. The ultimate goal of this pilot study is to identify feasible and potentially effective substance use stigma reduction interventions that go beyond simple individual-level professional training and that could be tested in a larger subsequent trial study.

This project will use a community-engaged approach with federally-qualified health centers (FQHCs) and other primary care sites to generate pilot data and establish protocols that not only measure self-reported changes in attitudes among health professionals but also use patient surveys and electronic medical records to measure the effect of educational and policy interventions on changes to clinical practice and patient outcomes.

Initial planning will focus on developing and pilot testing an educational curriculum (Aim 1) that addresses key drivers of provider-based stigma and FQHC facility recruitment and participation in policy development to address structural stigma (Aim 2). The latter half of the planning process will focus on refining and finalizing the trial design, survey instruments, data collection and management procedures, and drafting the trial protocol (Aim 3).

For Aim 1, the project team will design a curriculum addressing stigma related to substance use among the primary care workforce. The study team will prepare a 2-hour interactive curriculum to be used in an education session for individuals in any professional role (providers, other clinical support staff, and receptionists). The lead PI, Dr. Madden, will co-teach the course with a community consultant who has firsthand experience with SUD and harm reduction work. Including a co-teacher with such firsthand experience provides a contact-based approach to reducing stigma, which has been shown to reduce stigmatizing professional attitudes in several past studies. The curriculum will be piloted with ~35 primary care professionals, including physicians, other clinical support staff, and reception staff to assess changes to attitudes and intended behaviors that are indicative of substance use stigma. These changes will be assessed using validated surveys of provider-based stigma and new survey measures using the Theory of Planned Behavior to assess factors influencing professional behavior. A focus group with 6-10 pilot participants will be used to obtain qualitative feedback on the curriculum in order to refine and revise the training for the subsequent trial. The focus group will follow a Qualitative Description Approach, a methodology used in health services research to explore perspectives and experiences among people directly involved in a health/social phenomenon.

For Aim 2, FQHCs and other primary care sites providing HIV prevention and care services will be identified and approached in year 1 by the PIs. PIs will meet with interested FQHC administrators to explain the trial planning project and those administrators who agree to participate in trial planning will be asked to allow administrators and personnel to volunteer for qualitative interviews regarding facility policies and practices affecting stigma and HIV prevention and care for people who use drugs. In-depth semi-structured interviews with 15-20 FQHC professionals will be conducted in order to identify a suitable stigma policy to test in a larger subsequent trial study. Interviews will also be guided by the Qualitative Description Approach. Analyses will occur simultaneously with data collection and use thematic analysis. A policy proposal based on the qualitative analysis will be provided to FQHCs, and revised based on their feedback.

For Aim 3, the study team will collaborate with designated representatives ("champions") from each primary care site to design and finalize a trial protocol that tests a multi-level stigma intervention combining professional education and policy changes aimed at stigma reduction. The study team will work with the site champions in quarterly or monthly meetings (depending on scheduling availability of the champions) to review results from the training surveys, focus groups, and policy interviews, and to assure protocol feasibility and that site feedback is integrated into the pilot study and the ultimate goal of planning a larger subsequent trial study plans. A draft of the trial protocol will be provided to FQHC personnel along with anonymous online surveys soliciting feedback. The feedback will be analyzed by the project team and the organizational project champions, and the protocol will be revised.

The initial plan for the larger trial study that this pilot trial will inform includes a cluster randomized trial with 8 primary care sites and 80 primary care providers. Primary care providers will be the primary sampling units (i.e., the clusters), and patients will be the secondary sampling units. Randomization will first happen at the FQHC level so that all providers at a facility receive the same intervention in one of four arms: 1) facilities where personnel receive an educational intervention addressing provider-based stigma and facilities implement policy change aimed at reducing structural stigma toward PWUD; 2) facilities where personnel receive an educational intervention, but do not alter policies; 3) facilities that implement policy change, but personnel do not receive an educational intervention; and 4) control facilities without intervention implementation. For 20 random providers, 20 patients with substance use disorders (~400 patients total) will be selected in a second stage of randomization for survey participation. Patient surveys will include validated measures of anticipated, received, and internalized stigma, as well as validated tools to assess treatment adherence and use of harm reduction and substance use treatment services. Aggregated de-identified electronic medical records data from all patients of all participating providers will also be assessed as secondary sampling units. These patient outcomes for each primary care provider will be assessed to determine the effect of the multi-level stigma intervention. Electronic medical records and survey data will be collected for all arms at baseline and every 6 months for 24 months. Other clinical staff (e.g., nurses) and reception staff who interact with patients will be included in educational interventions, and may too be affected by policy changes (to be determined by outcomes of Aim 2), but will not be a primary sampling unit. The trial will require a separate IRB approval, and the current IRB approval is only for the pilot trial and planning activities in the R34.

ELIGIBILITY:
Inclusion Criteria:

* Employed at a federally qualified health center (FQHC) or other primary care site
* For training and focus group participants (primary outcomes), volunteer is involved in direct interaction with patients
* For interview and trial feasibility survey participants (secondary outcomes), volunteer is a decision-maker at the FQHC and/or directly interacts with patients

Exclusion Criteria:

* Not formally employed at a primary care facility (e.g., volunteer position at the site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the pilot training survey data or the qualitative interview data about the stigma policies.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from January 2023 - May 2023. Primary care professionals at two Michigan primary care sites were emailed information on the voluntary stigma training by site leadership and volunteers were solicited for responding to the pre-training and post-training surveys.
Pre-assignment Details: No volunteers were excluded form the study. All primary care professionals who volunteered were admitted to the training and allowed to participate in the surveys.
Period: Overall Study
Arm/Group | Training Group
Started | 51
Completed | 38
Not Completed | 13
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Population: Primary care providers currently employed at one of two Michigan federally qualified health centers
Arm/Group | Training Group
Number analyzed (Participants) | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51
job type [Count of Participants; unit: Participants]
  provider | 10
  clinic support staff (nurse, medical assistant) | 16
  Reception | 13
  Other staff | 12
site [Count of Participants; unit: Participants] — Which of two participating primary care sites the participants worked at
  Participants
    Primary care site 1 | 23
    Primary care site 2 | 28
burnout [Mean (Standard Deviation); unit: units on a scale] — "Overall, based on your definition of burnout, how would you rate your level of burnout?" 1= less burnout to 5= most burnout
  units on a scale | 2.04 (0.78)
past 3-month engagement with people who use drugs [Mean (Standard Deviation); unit: units on a scale] — 1= strongly disagree (Q: has engaged patients who use drugs and helped them to get evidence-based services) 5= strongly agree (Q: has engaged patients who use drugs and helped them to get evidence-based services)
  units on a scale | 2.92 (1.42)
Age, Customized [Count of Participants; unit: Participants] — age data not collected Population: age data not collected

OUTCOME MEASURES:

1. Primary Outcome: Provider-based Stigma (Social Distance Scale (SDS) Measure)
Description: This measure assesses how much "social distance" (level of contact/closeness they would prefer in social situations) that a respondent wants to have from a group of people. Four items from the social distance scale (SDS) adapted to people who use drugs. As reported in surveys taken by primary care professionals. Higher score= less social distance and less stigma. Minimum score on each SDS scale= 4; maximum score= 20. The intervention sought to promote higher scores (less desire for social distance, less stigma).
Time Frame: Change from baseline SDS score (measured 0-28 days prior to training) at 0-7 days post-training (pre/post design)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Training Group
Number analyzed (Participants) | 38
score on a scale
  pre-training mean SDS for people who currently use drugs | 9.09 [8.06 to 10.12]
  post-training mean SDS for people who currently use drugs | 11.89 [10.78 to 13.00]
Statistical Analysis 1: Comparison: Training Group; Test type: Other; p < 0.001, t-test, 2 sided

2. Primary Outcome: Provider-based Stigma (Medical Condition Regard Scale (MCRS) Measure)
Description: This measure assesses how positively healthcare professionals perceive a group of patients. Items from the Medical condition regard scale (MCRS) were adapted to patients who use drugs. As reported in surveys taken by primary care professionals. Higher score= more acceptance of the patient and lower stigma. Minimum score=7; maximum score=35. The intervention sought to promote higher scores (more acceptance, less stigma).
Time Frame: Change from baseline MCRS score (measured 0-28 days prior to training) at 0-7 days post-training (pre/post design)
Population: Primary care staff volunteers who attended the stigma training
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Training Group
Number analyzed (Participants) | 38
score on a scale
  Pre-training mean MCRS score | 22.70 [21.42 to 23.99]
  Post-training mean MCRS score | 25.03 [23.71 to 26.35]
Statistical Analysis 1: Comparison: Training Group; Test type: Other; p = 0.007, t-test, 2 sided

3. Primary Outcome: Provider-based Stigma (Planned Behavior Measure Assessing Intention to Help Patients Who Use Drugs)
Description: This measure used a single questions asking their level of agreement with the statement, "I intend to engage with patients who use drugs and help them to get evidence-based services over the next 3 months." This was reported in surveys taken by primary care professionals to assess planned stigmatizing actions based on the Theory of Planned Behavior. Higher score= more intention to help people who use drugs and less stigma. Maximum value=5; minimum value=1. The intervention sought to promote higher scores (more intention to help).
Time Frame: Change from baseline planned behavior score (measured 0-7 days prior to training) at 0-7 days post-training (pre/post design)
Population: primary care staff who volunteered to attend the training
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Training Group
Number analyzed (Participants) | 38
score on a scale
  Pre-training intention to help people who use drugs | 3.19 [2.82 to 3.55]
  Post-training intention to help people who use drugs | 3.57 [3.15 to 3.99]
Statistical Analysis 1: Comparison: Training Group; Test type: Other; p = 0.136, t-test, 2 sided

4. Primary Outcome: Number of Participants Who Completed Focus Groups on Training Feasibility
Description: The feasibility of the training was qualitatively assessed in focus groups using verbal feedback from participants. There was no quantification of this outcome other than counting how many participants provided feedback in the focus groups, and instead the feasibility of the training was assessed using thematic analysis, in which verbatim transcripts are read through and assigned brief analytic "codes" that briefly qualitatively summarize the content of participant feedback.
Time Frame: up to 5 months after the training
Population: Two nurses, two medical assistants, and one receptionist
Measure: Count of Participants; unit: Participants
Arm/Group | Training Group
Number analyzed (Participants) | 5
Participants | 5

5. Secondary Outcome: Number of Participants Who Completed Qualitative Interviews on Policy Feasibility
Description: Qualitatively assessed in in-depth interviews with primary care personnel. There was no quantification of this outcome other than counting how many participants provided feedback in the interviews, and instead the feasibility of the training was assessed using thematic analysis, in which verbatim transcripts are read through and assigned brief analytic "codes" that briefly qualitatively summarize the content of participant feedback.
Time Frame: One-time interview lasting 45-60 minutes per participant
Population: n=6 primary care providers, n=5 medical assistants, n=2 nurses, n=2 receptionists, n=2 senior administrators, n=4 other primary care staff
Measure: Count of Participants; unit: Participants
Arm/Group | Training Group
Number analyzed (Participants) | 21
Participants | 21

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Training Group
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT05925374/Prot_SAP_000.pdf